CLINICAL TRIAL: NCT02182570
Title: Phase III Open-labeled Study of WAL 801 CL Dry Syrup in Pediatric Atopic Dermatitis Patients
Brief Title: WAL 801 CL Dry Syrup in Pediatric Atopic Dermatitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 262.260
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

ARMS (1):
- WAL 801 CL (Experimental)
  Interventions: Drug: WAL 801 CL dry syrup

INTERVENTIONS:
Drug: WAL 801 CL dry syrup

SUMMARY:
The safety and efficacy of WAL 801 CL (epinastine hydrochloride) Dry Syrup in the treatment of atopic dermatitis in children was evaluated and plasma drug concentrations were measured.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in this study, subjects must be pediatric atopic dermatitis patients that meet the following criteria and thus be appropriate for observation of pruritus. Diagnosis of atopic dermatitis will be conducted in accordance with the "Definition and Diagnostic Criteria of Atopic Dermatitis", issued by the Japanese Dermatological Association.

* 15 years of age or younger
* Body weight of 14 kg or more
* Outpatients
* The patient has been undergoing treatment with a "very strong" or lower-grade external steroid preparation for >= 1 week at the time informed consent is obtained
* Pruritus with "2" or higher grade at the start time of administration

Exclusion Criteria:

* Use of sustained release adrenocorticotropic hormone (Kenacort® A, Depo-medrol®, etc.), oral preparation of methotrexate, or oral preparation of ciclosporin, within 4 weeks before initial administration of the investigational product
* Oral intake, inhalation and injection of any steroid within 2 weeks before initial administration of the investigational product
* Use of any external steroid preparation at "Strongest" in any sites other than the face or scalp within 2 weeks before initial administration of the investigational product
* Undergoing phototherapy
* Undergoing specific desensitization therapy or modulation therapy
* Past history of contact dermatitis caused by external steroid preparation
* Possibility of exacerbation by an external steroid preparation of infectious skin disease caused by bacteria, fungi, or virus
* Clinically significant hepatic, renal, or cardiac disease or other complications: therefore, judgement that the patient was ineligible for inclusion in this study. Patients must be excluded from the study if the patients fell under Grade 2 or more, in the MHW (Ministry of health and welfare) Adverse Reaction Severity Classification Criteria
* Past history of allergy to any drug
* Participation in any other clinical study, or history of participation in any other clinical study within 6 months before the date when the patient gave consent to participate in this study
* Judgement by the Principal Investigator or Investigator that the patient is ineligible for inclusion in this study

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2001-06; Primary Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Overall incidence of adverse events | up to 12 weeks
Occurrence of abnormal changes in laboratory measurements (haematological tests, blood biochemical tests, and urinalysis) | Baseline, weeks 4, 8 and 12

SECONDARY OUTCOMES:
Degree of pruritus | at weeks 4, 8 and 12
Degree of rash | at weeks 4, 8 and 12
Pruritus score obtained through the itching questionnaire | at weeks 4, 8 and 12
Impression on pruritus of the patient or the parent | week 12
Plasma concentration of epinastine hydrochloride | pre-dose and 6, 12, 18, 24, 30, 36 hours post-dose